CLINICAL TRIAL: NCT07270081
Title: Follicular Flushing Using Double Lumen Needle Versus Direct Aspiration in Low Prognosis Patients According to the POSEIDON Criteria
Acronym: FLUSHING
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto Bernabeu (Other)
Responsible Party: Principal Investigator, Dr. Paolo Cirillo, principal investigator, Instituto Bernabeu
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MR47
Record Dates: First submitted 2025-11-17; First posted 2025-12-08 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Low Ovarian Reserve; Poor Response to Ovulation Induction Poseidon Type IV; Poor Response to Ovulation Induction
Keywords: Follicular flushing; Poseidon 3 and 4; Poor responder; low ovarian reserve

STUDY DESIGN:
Intervention Model Description: Each participant will serve as her own control. One ovary will be randomized to single aspiration and the contralateral ovary to follicular flushing.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single Aspiration Arm (Active Comparator): Oocytes will be retrieved from one ovary using single follicular aspiration
  Interventions: Procedure: follicular aspiration
- Follicular Flushing Arm (Experimental): Oocytes will be retrieved from the contralateral ovary using follicular flushing, with up to three flushes per follicle if no cumulus-oocyte complex is obtained initially
  Interventions: Procedure: follicular flushing

INTERVENTIONS:
Procedure: follicular flushing — Follicles will be aspirated using 17G needles of the same gauge in both groups. For follicular flushing, the same type of needle used for single aspiration (Cook) will be employed. To eliminate dead space, the needle will be prefilled with flushing medium before starting the procedure. Aspiration pressure will be maintained at 190 mmHg during oocyte retrieval. In the follicular flushing group, if no cumulus-oocyte complex (COC) is recovered during the initial aspiration, follicular flushing will be performed until a COC is obtained, up to a maximum of three times. After three flushes, if no COC is retrieved, the procedure will be completed by rinsing with flushing medium to minimize the possibility of oocyte retention within the needle.
  Arms: Follicular Flushing Arm
Procedure: follicular aspiration — In the single aspiration group, after aspirating all follicles, the needle will be rinsed with flushing medium to prevent the possibility of oocyte retention within the needle.
  Arms: Single Aspiration Arm

SUMMARY:
This is a prospective, randomized, controlled clinical trial designed to evaluate whether follicular flushing increases the number of cumulus-oocyte complexes (COCs) retrieved compared to single aspiration in patients with poor ovarian response belonging to Poseidon groups 3 and 4.

A total of 40 patients with poor ovarian response belonging to Poseidon groups 3 and 4 will be included. In each patient, one ovary will be randomized to the study technique (follicular flushing), and the other ovary will be randomized to the control technique (single aspiration).

DETAILED DESCRIPTION:
This is a prospective, randomized, controlled clinical study designed to evaluate the effect of follicular flushing on the number of cumulus-oocyte complexes (COCs) retrieved, compared to single aspiration, in patients with poor ovarian response classified as Poseidon groups 3 and 4.

A total of 40 patients will be included. All participants will receive a standardized stimulation protocol consistent with current practice for patients diagnosed with low ovarian reserve. After meeting all inclusion criteria, controlled ovarian stimulation will begin within the first four days of the menstrual cycle, using an antagonist protocol in all cases.

Starting on the 6th day of ovarian stimulation, daily administration of a GnRH antagonist at a dose of 0.25 mg (Ganirelix® or Cetrorelix®) will be initiated. Final oocyte maturation will be triggered once at least one follicle reaches a diameter of ≥17 mm, using either 250 μg of recombinant hCG (Ovitrelle®; Merck Serono) or 0.2 mg of triptorelin acetate (Decapeptyl®), or a double trigger. Oocyte retrieval will be performed 36 hours after triggering final oocyte maturation.

On the day of oocyte retrieval, randomization will be performed using a computer-generated randomization list. In each patient, one ovary will be randomly assigned to the control group (single aspiration), and the contralateral ovary will be assigned to the study group (follicular flushing). Simple random allocation will be used. Each patient will be allowed to participate in the study only once.

Oocyte retrieval procedures will be performed by four trained physicians to evaluate the reproducibility and generalizability of the technique. Follicles will be aspirated using 17G needles in both groups. For follicular flushing, the same needle model used for single aspiration (Cook) will be employed. To eliminate dead space, the needle will be prefilled with flushing medium before beginning the procedure. Aspiration pressure will be maintained at 190 mmHg during oocyte retrieval.

In the single aspiration group, after aspirating all follicles, the needle will be rinsed with flushing medium to minimize the risk of oocyte retention inside the needle.

In the follicular flushing group, if no cumulus-oocyte complex (COC) is recovered during the initial aspiration, follicular flushing will be repeated until a COC is obtained, up to a maximum of three flushes. After three flushes, if no COC is retrieved, the procedure will be completed by rinsing with flushing medium to prevent possible oocyte retention within the needle.

The embryologist will immediately inform the physician performing the oocyte retrieval whether a COC has been recovered, in order to determine whether to continue flushing or proceed to the next follicle (open flushing technique).

The duration of the procedure will be recorded from needle insertion to its withdrawal for each ovary in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Pacientes con baja respuesta ovárica grupos POSEIDON 3 y 4 (< 35 años y RFA <5 y/o AMH < 1.2 ng/ml o > 35 años≥ 35 años y RFA <5 o AMH <1.2 ng/mL respectivamente)

  1. Pacientes menores o igual a 43 años.
  2. Índice de Masa Corporal (IMC) de 18-35 kg/m2
  3. Estimulación ovárica para ICSI
  4. Presencia y accesibilidad de ambos ovarios.
  5. Ausencia de patología ovárica
  6. Cuando se cumplan los criterios de desencadenamiento para la maduración final del ovocito, cada ovario debe contener al menos un folículo mayor o igual a 14 mm.
  7. Haber dado su consentimiento por escrito.

Exclusion Criteria:

* Presence of a single ovary.

Presence of ovarian pathology.

Use of conventional IVF as the fertilization method.

Max Age: 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
number of cumulus-oocyte complexes | During the egg retrieval
  number of cumulus-oocyte complexes (COCs) retrieved after each aspiration

SECONDARY OUTCOMES:
Oocyte recovery rate | day of the egg retrieval
  number of oocytes retrieved / number of follicles ≥11 mm on the day of final oocyte maturation trigger
Fertilization rate | 1 day after the egg retrieval
  number of 2PNs / number of MII oocytes
Empty follicle rate | day of the egg retrieval
  zero oocytes retrieved / follicles punctured
Procedure time | In seconds from needle insertion to its withdrawal for each ovary
  calculated from needle insertion to its withdrawal for each ovary

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Bernabeu, Alicante, Alicante, Spain

IPD SHARING:
Plan to Share IPD: Undecided